CLINICAL TRIAL: NCT05158673
Title: Effect of Cocoa Polyphenols Supplementation on Cardiovascular Risk of Overweight or Obese Postmenopausal Women: Double Blind Randomized Clinical Trial
Brief Title: Effect of Cocoa Polyphenols Supplementation on Cardiovascular Risk of Postmenopausal Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes (Other Government)
Collaborators: National Polytechnic Institute, Mexico (Other)
Responsible Party: Principal Investigator, Araceli Montoya-Estrada, Clinical Researcher, Instituto Nacional de Perinatologia Isidro Espinosa de los Reyes
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-1-29
Record Dates: First submitted 2021-11-17; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Metabolic Syndrome
Keywords: flavonoids; cocoa; postmenopausal women; metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized Clinical Trial only the principal investigator is not blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Placebo) (Placebo Comparator): The administration of two capsules of 500 mg orally of placebo (excipient q.s. starch capsule) 1 every 12 hours, for 12 weeks.
  Interventions: Dietary Supplement: Placebo of Cocoa flavonoids
- Group B (Flavonoid) (Active Comparator): Two capsules of 500 mg of the flavonoid supplement (whose total flavonoid content is 15 mg/capsule) orally every 12 hours for 12 weeks.
  Interventions: Dietary Supplement: Cocoa flavonoids

INTERVENTIONS:
Dietary Supplement: Placebo of Cocoa flavonoids — Dietary supplement: The administration of two capsules of 500 mg orally of placebo (excipient q.s. starch capsule) 1 every 12 hours, for 12 weeks
  Arms: Group A (Placebo)
Dietary Supplement: Cocoa flavonoids — Dietary supplement: Two 500 mg capsules of the flavonoid supplement (whose total flavonoid content is 15 mg/capsule) orally every 12 hours (one in the morning and one at night) for 12 weeks
  Arms: Group B (Flavonoid)

SUMMARY:
Several epidemiological studies have shown that premenopausal women are protected from cardiovascular diseases compared to men of the same age; however, after menopause (postmenopause), the cardiovascular risk increases progressively to equal the cardiovascular risk of men of the same age group. In addition, in Mexico, the incidence of women entering the postmenopausal stage with overweight or obesity increases each year. Therefore, it is essential to generate public initiatives to reduce the metabolic and physiological alterations caused by overweight/obesity and improve postmenopausal women's health and quality of life. Flavonoids are bioactive compounds that have been shown to reduce the cardiovascular risk associated with obesity since they participate in the regulation of lipid metabolism, improve body composition, reduce oxidative stress and inflammation; Therefore, our objective is to reduce the cardiovascular risk of postmenopausal women and improve the oxidative and inflammatory state, through oral supplementation with cocoa flavonoids. To do this, an innovative method will be used to assess cardiovascular risk based on knowledge of the type, number, and size of lipoprotein particles and knowing the oxidative and inflammatory state before and after supplementation with cocoa flavonoids.

DETAILED DESCRIPTION:
Some interventions have been carried out to reduce obesity and the incidence of cardio-metabolic pathologies since the foods consumed in the daily diet, directly and indirectly, influence the modulation of metabolic signaling pathways. Flavonoids, nutrients of plant origin, have beneficial effects on health since they can prevent and reduce the impact of overweight/obesity. Significant benefits have also been shown in blood pressure, platelet reactivity, HDL cholesterol, LDL cholesterol, insulin sensitivity, and prostaglandin metabolism, improving health in patients with chronic diseases related to metabolic disorders and OS.

Food rich in flavonoids is cocoa; the plant contains many polyphenols (anthocyanidins, proanthocyanidins, and catechins), concentrated mainly in the pods and seeds, which provides a highly bitter taste. The polyphenols that can be identified in cocoa beans are (-) - epicatechin and, to a lesser extent (+) - catechin, (+) - gallocatechin, and (-) - epigallocatechin.

Polyphenols derived from cocoa are characterized by being powerful antioxidants, by having effects on muscle and fat tissue: inducing the darkening of adipocytes (change from white adipocytes (fat deposit) to beige adipocytes; promoting mitochondrial biogenesis; increasing the expression of vital thermogenic genes and upstream regulators of fatty acid oxidation; reducing serum TG concentrations; phosphorylating metabolism regulators and acetylating (activating) proteins involved in mitochondrial structure and function. Actions culminate in regulating the metabolic profile, decreasing adipose tissue, increasing muscle mass, and, therefore, decreasing BMI.

There is evidence of the beneficial effects of cocoa polyphenols as antioxidants, improving the lipid profile levels and pro and anti-inflammatory markers. Cocoa is one of the foods of natural origin with high antioxidant capacity due to the tricyclic structure of flavonoids. The compounds act as electron donors and stabilize free radicals through their aromatic rings with hydroxyl substituents. Cocoa polyphenols have been shown to protect cells from oxidative stress at the membrane level by reducing lipoperoxidation and DNA damage through the chelating action of the catechol group and hydroxyl substituents. Furthermore, cocoa flavonoids inhibit xanthine oxidase, NADPH-oxidase, tyrosine kinases, and protein kinases.

Cocoa polyphenols have been shown to have antioxidant activity that helps counteract the atherosclerotic process by reducing the activation of NADPH oxidase. In addition, to improve the dilation of the arteries in smoking patients with atherosclerosis. The antioxidants in cocoa inhibit LDL oxidation, which is related to delaying atherosclerotic progression by reducing ox-LDL and increasing HDL-c.

ELIGIBILITY:
Inclusion Criteria:

* -According to the STRAW classification (+ 1A + 1B + 1C), women with an early postmenopause diagnosis attend the INPerIER Peri and Postmenopause Clinic.
* Age between 50 and 60 years.
* who have metabolic syndrome
* Who present an altered lipid and glycemic profile that have not reached the critical point of pharmacological treatment (blood glucose between 100 and 125 mg/dl, cholesterol between 200 and 280 mg/dl, triglycerides between 150 and 300 mg/dl, lower HDL 50 mg/dl).
* That they are not taking metformin
* That they have not taken metformin in the three months before entering the study.
* That they are not taking bezafibrate and/or statins.
* That they have not taken bezafibrate and/or statins in the three months before entering the study.
* No indication for hormone replacement therapy.
* That they sign the informed consent.

Exclusion Criteria:

* Women who present pathologies such as Diabetes Mellitus, rheumatoid arthritis, lupus, neoplasms of any type, HIV, or kidney diseases during the development of the study.
* Women who require hormone replacement therapy during the development of the protocol.
* That the patient has any surgical intervention during the development of the study.
* Women who consume or require the use of lipid-lowering drugs during the development of the protocol

Ages: 50 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women with an early postmenopause diagnosis
Enrollment: 30 (Estimated)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Metabolic Syndrome | Metabolic Syndrome at three months after starting the intervention in each group
  Metabolic syndrome according to International Diabetes Federation Criteria

SECONDARY OUTCOMES:
Carbonylation of proteins | Three months after starting the intervention in each group
  Marker of oxidative stress measured by spectrophotometry expressed as pmol PC/mg protein
Malondialdehyde | Three months after starting the intervention in each group
  Marker of oxidative stress measured by spectrophotometry expressed as pmol MDA/mg dry weight
Superoxide Dismutase activity | Three months after starting the intervention in each group
  Enzymatic activity measured by Colorimetric Activity Kit expressed as nmol/min/mL
Catalase activity | Three months after starting the intervention in each group
  Enzymatic activity measured by Colorimetric Activity Kit expressed as nmol/min/mL
Lipid profile quantification | Three months after starting the intervention in each group
  size of cholesterol (main classes and subclasses of lipoproteins) expressed in large, medium and small)
IL-4, IL-6, IL10 and TNFa | Three months after starting the intervention in each group
  They will be quantified by ELISA technique expressed in pg/ul

CONTACTS AND LOCATIONS:
Overall Officials: Araceli Montoya-Estrada, PhD, Principal Investigator — Instituto Nacional de Perinatología Isidro Espinosa de los Reyes; Nayelli Najera, PhD, Study Director — Instituto Politecnico Nacional
Locations (1):
- Instituto Nacional de Perinatología Isidro Espinosa de los Reyes, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
no applicable

REFERENCES:
- [Background] Goya L, Martin MA, Sarria B, Ramos S, Mateos R, Bravo L. Effect of Cocoa and Its Flavonoids on Biomarkers of Inflammation: Studies of Cell Culture, Animals and Humans. Nutrients. 2016 Apr 9;8(4):212. doi: 10.3390/nu8040212. PMID 27070643
- [Background] Gutierrez-Salmean G, Meaney E, Lanaspa MA, Cicerchi C, Johnson RJ, Dugar S, Taub P, Ramirez-Sanchez I, Villarreal F, Schreiner G, Ceballos G. A randomized, placebo-controlled, double-blind study on the effects of (-)-epicatechin on the triglyceride/HDLc ratio and cardiometabolic profile of subjects with hypertriglyceridemia: Unique in vitro effects. Int J Cardiol. 2016 Nov 15;223:500-506. doi: 10.1016/j.ijcard.2016.08.158. Epub 2016 Aug 8. PMID 27552564